CLINICAL TRIAL: NCT06197802
Title: An Observational Study to Compare Plateau Antibody Levels of a Recombinant (E.Coli) Human Papillomavirus Nonavalent (Type 6/11/16/18/31/33/45/52/58) Vaccine Versus Gardasil®9 in Healthy Females 18-26 Years of Age
Brief Title: Plateau Antibody Levels of a Recombinant (E.Coli) HPV Nonavalent Vaccine Versus Gardasil®9 in Young Women
Status: Active, not recruiting | Type: Observational
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Other Study IDs: HPV-PRO-011-1
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; Condylomata Acuminata
Keywords: human papillomavirus vaccine
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58) Vaccine(E.Coli) group: Subjects would receive 3 doses of 270μg/0.5ml Recombinant HPV nonavalent (Types 6/11/16/18/31/33/45/52/58) Vaccine(E.Coli)
  Interventions: Biological: Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58 )Vaccine(E.Coli)
- Gardasil®9 group: Subjects would receive 3 doses of 270μg/0.5ml Gardasil®9
  Interventions: Biological: Gardasil®9

INTERVENTIONS:
Biological: Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58 )Vaccine(E.Coli) — Three doses administered intramuscularly at 0, 45 day and 6 month.
  Groups: Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58) Vaccine(E.Coli) group
Biological: Gardasil®9 — Three doses administered intramuscularly at 0, 45 day and 6 month.
  Groups: Gardasil®9 group

SUMMARY:
This study is designed to compare plateau antibody levels of a novel recombinant human papillomavirus vaccine (types 6,11,16,18,31,33,45,52,58 )(E.Coli) manufactured by Xiamen Innovax Biotech CO., Ltd., with Gardasil®9 in females 18-26 Years of Age.

ELIGIBILITY:
Inclusion Criteria:

* Subject who had previously participated in the Randomized, Single-blind Study to Compare Immunogenicity of a Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58) Vaccine(E.Coli) (Xiamen Innovax Biotech Co.,Ltd.) Versus Gardasil®9 (Merck & Co., Inc.) in Healthy Females 18-26 Years of Age (Protocol No.: HPV-PRO-011, Identifiers: NCT04782895), and received at least one dose ;
* Subject is able to understand and comply with the requirements of the protocol(e.g. biological specimen collection, return for follow-up visits), and written informed consent must be obtained from the subject prior to enrollment;

Exclusion Criteria:

* Subject who had used other HPV vaccine products (including marketed and unmarketed vaccines) after participating in the Randomized, Single-blind Study to Compare Immunogenicity of a Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58) Vaccine(E.Coli) (Xiamen Innovax Biotech Co.,Ltd.) Versus Gardasil®9 (Merck & Co., Inc.) in Healthy Females 18-26 Years of Age (Protocol No.: HPV-PRO-011, Identifiers: NCT04782895) ;
* Subject has abnormal coagulation function (such as coagulation factor deficiency, coagulopathy, platelet abnormalities) or coagulation disorders;
* Medical, psychological, social conditions, occupation or other factors, which considered by the investigator that may influence the conduct of the clinical study.

Ages: 20 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subject who had previously participated in the Randomized, Single-blind Study to Compare Immunogenicity of a Recombinant Human Papillomavirus Nonavalent (Types 6,11,16,18,31,33,45,52,58) Vaccine(E.Coli) (Xiamen Innovax Biotech Co.,Ltd.) Versus Gardasil®9 (Merck & Co., Inc.) in Healthy Females 18-26 Years of Age (Protocol No.: HPV-PRO-011, Identifiers: NCT04782895), and received at least one dose
Sampling Method: Non-Probability Sample
Enrollment: 392 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 type specific neutralizing antibody level | 30-36 months after the first dose
  Anti-HPV 6,11,16,18,31,33,45,52 and 58 seropositive rates and geometric mean concentrations at months 30-36

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, master, Study Chair — Xiamen University; Feng-cai Zhu, master, Principal Investigator — Jiangsu Provincial Centre for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Centre for Disease Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhong GH, Bi ZF, Chu K, Zhang L, Chen L, Zhu KX, Quan JL, Nie C, Chen Q, Qiu LX, Xu JB, Li JX, Zhang ML, Liu S, Nie LL, Li K, Su YY, Huang SJ, Zhang QF, Huang WJ, Pan HX, Wu T, Zhang J, Xia NS. Immunogenicity comparison of an Escherichia coli-produced 9-valent human papillomavirus vaccine and Gardasil9 in Chinese women aged 18-26 years: three-year follow-up data from a randomised clinical trial. Lancet Reg Health West Pac. 2025 Aug 27;62:101671. doi: 10.1016/j.lanwpc.2025.101671. eCollection 2025 Sep. PMID 40919385